CLINICAL TRIAL: NCT04219111
Title: Detecting Expression Profiles Associated With Resistance to Tyrosine Kinase Inhibitors in Chronic Myeloid Leukaemia Patients Without Detectable Tyrosine Kinase Domain Mutations, Using Transcriptomics
Brief Title: Gene Expression Profiles in CML Non-responders
Status: Withdrawn | Type: Observational
Why Stopped: STUDY LOOKING AT SAMPLES ONLY, NO PARTICIPANT ENROLMENT REQUIRED
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SCH-2181
Record Dates: First submitted 2020-01-03; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Gene Expression Profiles in CML Non-responders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Using retrospective anonymised DNA samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Clariom — Clariom S Assay

SUMMARY:
Chronic myeloid leukaemia (CML) is a haematological malignancy primarily driven by the fusion oncogene BCR-ABL1, resulting in a constitutively expressed tyrosine kinase. CML is treated very effectively by the tyrosine kinase inhibitors (TKIs) resulting in almost undetectable levels of disease. However, some patients show resistance to first line treatment, requiring second and third generation TKIs. Such resistance is due to the presence of tyrosine kinase domain (TKD) mutations, however TKDs do not appear to be present in all patients who do not respond to treatment.

The aim of this project is to utilise gene expression arrays to identify transcriptomic profiles associated with resistance to TKIs in the absence of a demonstrable TKD mutation. The presence of such profiles may allow for a more targeted approach to treatment, if non-responders can be identified earlier in the disease management pathway. Being able to predict those that will not respond to first line treatment will allow for better stratification of patients.

DETAILED DESCRIPTION:
The aim of this project is to use gene expression microarrays to detect expression profiles which may be associated with TKI resistance in order to better stratify CML patients and allow a more targeted approach to therapy. The project may also help elucidate the mechanism of resistance in those without a discernible TKD mutation. Ultimately it is hoped that this would lead to larger studies which could improve the clinical pathway for CML patients without TKD mutations.

Some previous studies have studied the gene expression profile of CML patients demonstrating resistance to TKIs, using Affymetrix arrays. However, none of these appear to have specifically investigated non-responders with and without a TKD mutation.

ELIGIBILITY:
Inclusion Criteria:

* CML patients with poor response to TKIs as identified through routine clinical testing at SDGS, either with or without a tyrosine kinase domain mutation as tested for by mutational analysis.

Exclusion Criteria:

* Any samples that do not meet the above inclusion criteria, but particularly not CML patients with an optimal response to TKIs.

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CML patients with poor response to TKIs as identified through routine clinical testing at SDGS, either with or without a tyrosine kinase domain mutation as tested for by mutational analysis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Success identification of at least 5 markers of resistance in patients without a TKD mutation and confirmation of their expression levels using qPCR | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No